CLINICAL TRIAL: NCT03893253
Title: Does an Early Booster Session Improve Performance and Retention of Basic Life Support Skills Compared to a Late Booster in Health Care Professionals? A Simulation-based Randomized Controlled Trial.
Brief Title: Early or Late Booster in Basic Life Support for Health Care Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Collaborators: Institut du Savoir Montfort (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-19-08-020
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Basic Life Support

STUDY DESIGN:
Intervention Model Description: Participants randomized to one of three groups : early booster, late booster, or no booster (control group)
Who Masked: Outcomes Assessor
Masking Description: Trained evaluators will rate a series of videos but will be blinded to which arm of the study participants are from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Booster Teaching (Experimental): The early booster group will receive a booster teaching session at 3 weeks post-training followed by feedback.
  Interventions: Other: Early Booster Teaching
- Late Booster Teaching (Active Comparator): The late booster group will receive a booster teaching session at 2 months post-training followed by feedback.
  Interventions: Other: Late Booster Teaching
- Control group (No Intervention): The control group will receive no booster teaching at all.

INTERVENTIONS:
Other: Early Booster Teaching — The early booster group will receive a booster teaching session at 3 weeks post-training followed by feedback.
  Arms: Early Booster Teaching
Other: Late Booster Teaching — The late booster group will receive a booster teaching session at 2 months post-training followed by feedback
  Arms: Late Booster Teaching

SUMMARY:
Attrition of skills after basic life support (BLS) training is common. Psychology studies have established that for basic memory recall tasks, spaced learning strategies improve retention. Spaced learning is often organized as a refresher or 'booster' course after initial training. This study aims to investigate if this principle holds true for BLS skills, which require rapid memory recall and efficient deployment of procedural skills while under time pressure.

DETAILED DESCRIPTION:
Health care professionals who have not received BLS training in the 6 months leading up to the date of participation will be recruited from local health care institutions in the greater-Ottawa area. Participants will be randomized into one of three groups: early booster, late booster, or no booster (control). Currently, no booster is the educational standard. The early booster group will receive a booster at 3 weeks, the late booster at 2 months, and no booster for the control. All participants will undergo BLS training, an immediate post-test, and a retention post-test at 4 months. Post-tests involve a simulated cardiac arrest scenario. Raters will be blinded to the group allocation and simulation test order.

ELIGIBILITY:
Inclusion Criteria:

-Healthcare professionals who interact with patients and have not received any BLS training or practice in the 6 months leading up to the date of their participation will be recruited.

Exclusion Criteria:

* under 18 years of age
* non healthcare professionals
* healthcare professionals who don't interact directly with patients
* healthcare professionals who have completed Basic Life Support training in the previous six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Basic Life Support Performance | 4 months
  Basic Life Support performance, as measured by the standardized Heart and Stroke checklist score

SECONDARY OUTCOMES:
Time to start chest compressions | 4 months
  Time from entering the scene to initiation of compression
Time to defibrillation | 4 months
  Time from start to defibrillation with AED
Quality of CPR | 4 months
  Hand placement on lower half of sternum, 30 compressions in no less than 15 and no more than 18 seconds, compresses at least 5 cm, complete recoil after each compression
Overall BLS performance | 4 months
  Basic Life Support performance, as measured by the standardized Heart and Stroke checklist (PASS OR FAIL)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Waldolf, MD, Principal Investigator — Hôpital Montfort
Locations (1):
- Institut du Savoir Montfort, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No